CLINICAL TRIAL: NCT00641706
Title: Phase II Study of Vorinostat (SAHA) in Combination With Bortezomib (PS-341) in Patients With Recurrent Glioblastoma Multiforme
Brief Title: Vorinostat and Bortezomib in Treating Patients With Progressive, Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00668; NCI-2009-00668 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000590113; NCCTG-N0779; N0779 (Other: North Central Cancer Treatment Group); N0779 (Other: CTEP); U10CA025224 (NIH)
Record Dates: First submitted 2008-03-21; First posted 2008-03-24 (Estimated); Results first posted 2013-07-10 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2011-10

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Vorinostat; Bortezomib

ARMS (2):
- Stratum 1 (not undergoing surgery) (Experimental): Patients receive oral vorinostat (SAHA) once daily on days 1-14 and bortezomib IV on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vorinostat; Drug: bortezomib
- Stratum 2 (undergoing surgery) (Experimental): Patients receive oral SAHA once daily for 2 days prior to surgery and then on the day of surgery. Patients also receive bortezomib IV on the day of surgery. After receiving the 3rd dose of SAHA, patients undergo surgery to remove the tumor. Beginning at least 7 days after surgery, patients receive SAHA and bortezomib as in stratum 1.
  Interventions: Drug: vorinostat; Procedure: therapeutic conventional surgery; Drug: bortezomib

INTERVENTIONS:
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Procedure: therapeutic conventional surgery — Patient undergoes surgery
  Arms: Stratum 2 (undergoing surgery)
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE

SUMMARY:
This phase II trial is studying how well giving vorinostat together with bortezomib works in treating patients with progressive, recurrent glioblastoma multiforme. Vorinostat and bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving vorinostat together with bortezomib may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the clinical efficacy of vorinostat (SAHA) and bortezomib, in terms of progression-free survival (PFS) at 6 months, in patients with progressive, recurrent glioblastoma multiforme.

SECONDARY OBJECTIVES:

I. To determine the clinical efficacy of this regimen, in terms of overall survival, PFS at 12 months, time to progression, and objective response rate, in these patients.

II. To identify molecular predictors of response in baseline tumor specimens from these patients.

III. To determine molecular changes in response to this regimen in tumor specimens from patients undergoing surgery.

OUTLINE: This is a multicenter study. Patients are stratified according to planned surgery (no [stratum 1] vs yes [stratum 2]).

STRATUM 1 (NOT UNDERGOING SURGERY): Patients receive oral vorinostat (SAHA) once daily on days 1-14 and bortezomib intravenously (IV) on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

STRATUM 2 (UNDERGOING SURGERY): Patients receive oral SAHA once daily for 2 days prior to surgery and then on the day of surgery. Patients also receive bortezomib IV on the day of surgery. After receiving the 3rd dose of SAHA, patients undergo surgery to remove the tumor. Beginning at least 7 days after surgery, patients receive SAHA and bortezomib as in stratum 1.

Tumor tissue samples are collected at baseline and during surgery (stratum 2) for correlative laboratory studies. Tissue samples are analyzed for baseline total and phosphorylated AKT and p27^KIp1 expression by IHC. Tissue samples from patients in stratum 2 are also analyzed for histone acetylation status; markers of proteasome inhibition; total and phosphorylated Bax expression by IHC; and gene expression profiles.

After completion of study therapy, patients are followed every 3 months for 2 years and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed glioblastoma multiforme

  * Gliosarcoma or other grade 4 astrocytoma variant (e.g., giant cell glioblastoma) allowed
  * Recurrent disease
* Must have evidence of tumor progression by MRI or CT scan after radiotherapy or after the most recent antitumor therapy
* Bidimensionally measurable or evaluable disease by MRI or CT scan

  * Patients receiving corticosteroids must be on a fixed dose for at least 1 week prior to baseline scan
* ECOG performance status 0-2
* WBC ≥ 3,000/mm³
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST ≤ 3 times ULN
* Creatinine normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after the last dose of vorinostat
* Willing to provide mandatory correlative laboratory tissue samples
* Able to take oral medications
* No uncontrolled infection
* No known hypersensitivity to any of the components of vorinostat or bortezomib
* No myocardial infarction or unstable angina within the past 6 months
* No congestive heart failure requiring use of ongoing maintenance therapy or history of life-threatening ventricular arrhythmias
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Psychiatric illness or social situation that would limit compliance with study requirements
* No other active malignancy within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No comorbid systemic illness or other severe concurrent disease that, in the judgment of the investigator, would preclude study entry or significantly interfere with proper assessment of safety and toxicity of the prescribed study regimens
* Not immunocompromised

  * Patients known to be HIV positive are eligible provided there is no clinical evidence of an immunocompromised state
* No peripheral neuropathy ≥ grade 2
* No peripheral neuropathy with pain ≥ grade 1
* No congenital long QT syndrome
* No prolonged OTC interval (> 450 msec)
* No other concurrent anticancer therapy (other than hormonal therapy)
* At least 8 weeks since prior radiotherapy
* More than 6 weeks since prior stereotactic radiosurgery or interstitial brachytherapy, unless there is a separate lesion on MRI that is not part of the prior treatment field
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* No more than 1 prior chemotherapy regimen* for progressive/recurrent disease (stratum 1)

  * Patients in stratum 2 may have received any number of prior chemotherapy regimens* for progressive/recurrent disease
* More than 2 weeks since prior small molecule cell cycle inhibitors
* More than 7 days since prior valproic acid
* More than 7 days since prior category I drugs that are generally accepted to have a risk of causing Torsades de Pointes including:

  * Quinidine, procainamide, disopyramide
  * Amiodarone, sotalol, ibutilide, dofetilide
  * Erythromycin, clarithromycin
  * Chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide
  * Cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin,lidoflazine
* More than 4 weeks since prior bevacizumab
* No prior treatment with vorinostat or bortezomib
* No concurrent enzyme-inducing antiepileptic drugs (e.g., phenytoin,fosphenytoin, carbamazepine, phenobarbital, or primidone)
* No other concurrent potent CYP3A4 inducer (e.g., rifampin or St. John's wort)
* No other concurrent investigational therapy for the primary neoplasm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-07; Primary Completion 2010-07 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Galanis, Principal Investigator — North Central Cancer Treatment Group
Locations (214):
- United States (214):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Cottage, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Carle Clinic-Urbana Main, Urbana, Illinois
  - Saint Francis Hospital and Health Centers, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Cedar Rapids Oncology Association, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Mercy Health Partners-Hackley Campus, Muskegon, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Duluth Clinic CCOP, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies PC, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis HealthCare System, Zanesville, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - AnMed Health Hospital, Anderson, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Upstate Carolina CCOP, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Midelfort Clinic-Clairemont Campus, Eau Claire, Wisconsin
  - Mayo Clinic Health System Eau Claire Hospital - Luther Campus, Eau Claire, Wisconsin
  - Agnesian Cancer Center, Fond du Lac, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 45 patients were enrolled from 28 medical clinics between July 4, 2008 and February 16, 2010.
Pre-assignment Details: One patient cancelled prior to treatment initiation and is excluded in the analysis.
Groups:
- Arm A (Not Undergoing Surgery): Patients receive oral vorinostat (SAHA) once daily on days 1-14 and bortezomib IV on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  bortezomib : Given IV
  vorinostat : Given orally
- Arm B (Undergoing Surgery): Patients receive oral SAHA once daily for 2 days prior to surgery and then on the day of surgery. Patients also receive bortezomib IV on the day of surgery. After receiving the 3rd dose of SAHA, patients undergo surgery to remove the tumor. Beginning at least 7 days after surgery, patients receive SAHA and bortezomib as in stratum 1.
  surgery : Patient undergoes therapeutic conventional surgery
  bortezomib : Given IV
  vorinostat : Given orally
Period: Overall Study
Arm/Group | Arm A (Not Undergoing Surgery) | Arm B (Undergoing Surgery)
Started | 37 | 7
Completed | 28 | 4
Not Completed | 9 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Clinical Decline | 1 | 0
Not completed — Lead Investigator Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Not Undergoing Surgery) | Arm B (Undergoing Surgery) | Total
Number analyzed (Participants) | 37 | 7 | 44
Age, Continuous [Median (Full Range); unit: years] | 52 [33 to 80] | 51 [39 to 60] | 52 [33 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 1 | 11
  Male | 27 | 6 | 33
Region of Enrollment [Number; unit: participants]
  United States | 37 | 7 | 44

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 6 Months
Description: Estimated using the Binomial point estimator (number of successes divided by the total number of evaluable patients). A patient is classified as a success if alive and progression-free at 6 months. For patients with bidimensionally measurable disease (measurable disease), progression is defined as > 25% increase in product of perpendicular diameters of contrast enhancement or mass or appearance of new lesions. For patients without bidimensionally measurable disease (evaluable disease), progression is defined as unequivocal increase in size of contrast enhancement or increase in mass effect as agreed upon independently by primary physician and quality control physicians or appearance of new lesions.
Time Frame: At 6 months
Population: Patients that started treatment.
Measure: Number; unit: percentage of patients
Arm/Group | Arm A (Not Undergoing Surgery) | Arm B (Undergoing Surgery)
Number analyzed (Participants) | 37 | 7
percentage of patients | 0 | 29

2. Secondary Outcome: Overall Survival
Description: Estimated using Kaplan-Meier survival curve.
Time Frame: From study registration to date of death due to any cause or last follow-up (up to 5 years)
Population: Patients that started treatment.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A (Not Undergoing Surgery) | Arm B (Undergoing Surgery)
Number analyzed (Participants) | 37 | 7
months | 3.2 [0.7 to 24.8] | 8.7 [3.0 to 16.4]

3. Secondary Outcome: Time to Progression
Description: Estimated using Kaplan-Meier survival curve. Patients who died were considered to have disease progression at the time of death unless there was documented evidence that no progression occurred before death. For patients with bidimensionally measurable disease (measurable disease), progression is defined as > 25% increase in product of perpendicular diameters of contrast enhancement or mass or appearance of new lesions. For patients without bidimensionally measurable disease (evaluable disease), progression is defined as unequivocal increase in size of contrast enhancement or increase in mass effect as agreed upon independently by primary physician and quality control physicians or appearance of new lesions.
Time Frame: From study registration to date of progression (up to 5 years)
Population: Patients that started treatment.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A (Not Undergoing Surgery) | Arm B (Undergoing Surgery)
Number analyzed (Participants) | 37 | 7
months | 1.5 [0.5 to 5.6] | 4.2 [0.6 to 9.3]

4. Secondary Outcome: Proportion of Confirmed Tumor Response Defined as an Objective Status of Confirmed Response (CR), Partial Response (PR), or Regression (REGR) on Two Consecutive Evaluations
Description: Confidence intervals for the true proportion will be calculated using the exact binomial method.
  Measurable patients must achieve at least a 50% reduction in the product of perpendicular diameters of contrast enhancement or mass with no new lesions with the patient being on stable or decreased steroid dose.
  Evaluable patients must achieve unequivocal reduction in size of contrast-enhancement or decrease in mass effect as agreed upon independently by primary physician and quality control physicians; no new lesions. Patient should be on stable or decreased steroid dose.
Time Frame: Assessed up to 5 years
Population: Arm A patients that started treatment. Arm B patients were not analyzed for this outcome because they received surgery and hence response was not measured.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Arm A (Not Undergoing Surgery) | Arm B (Undergoing Surgery)
Number analyzed (Participants) | 37 | 0
proportion of patients | 0.027 [0.0007 to 0.14] |

ADVERSE EVENTS:
Groups:
- Arm A (Not Undergoing Surgery); Arm B (Undergoing Surgery): vorinostat : Given orally
Arm/Group | Arm A (Not Undergoing Surgery) | Arm B (Undergoing Surgery)
Serious Adverse Events (participants affected / at risk) | 18/37 | 0/7
Other Adverse Events (participants affected / at risk) | 36/37 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Not Undergoing Surgery) (N=37) | Arm B (Undergoing Surgery) (N=7)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Opportunistic infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 12 (13) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (2) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Personality change (Psychiatric disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Not Undergoing Surgery) (N=37) | Arm B (Undergoing Surgery) (N=7)
Hemoglobin decreased (Blood and lymphatic system disorders) | 23 (45) | 5 (6)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Dry eye syndrome (Eye disorders) | 0 (0) | 1 (3)
Vision blurred (Eye disorders) | 2 (4) | 0 (0)
Watering eyes (Eye disorders) | 2 (5) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 10 (16) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 9 (13) | 3 (6)
Dry mouth (Gastrointestinal disorders) | 2 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 4 (5) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 14 (24) | 4 (6)
Vomiting (Gastrointestinal disorders) | 8 (9) | 1 (1)
Edema limbs (General disorders) | 4 (7) | 0 (0)
Fatigue (General disorders) | 31 (70) | 5 (15)
Pain (General disorders) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 3 (8) | 0 (0)
Creatinine increased (Investigations) | 2 (2) | 0 (0)
Leukocyte count decreased (Investigations) | 11 (16) | 1 (2)
Lymphocyte count decreased (Investigations) | 5 (6) | 2 (3)
Neutrophil count decreased (Investigations) | 7 (7) | 1 (1)
Platelet count decreased (Investigations) | 31 (55) | 5 (11)
Weight gain (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 3 (3) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 8 (12) | 2 (3)
Blood glucose increased (Metabolism and nutrition disorders) | 4 (10) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 7 (8) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Serum potassium increased (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (7) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4)
Acoustic nerve disorder NOS (Nervous system disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 3 (3) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (2) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 5 (6) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Mini mental status examination abnormal (Nervous system disorders) | 2 (3) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (11) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 1 (1)
Speech disorder (Nervous system disorders) | 2 (3) | 0 (0)
Taste alteration (Nervous system disorders) | 5 (15) | 1 (1)
Confusion (Psychiatric disorders) | 2 (5) | 0 (0)
Depression (Psychiatric disorders) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (4) | 0 (0)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 0 (0)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (9) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (5) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (5) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less